CLINICAL TRIAL: NCT04241406
Title: Transcutaneous Spinal Cord Stimulation in Healthy Subjects to Activate Central Pattern Generator: Double-blind, Randomised, Controlled Clinical Trial.
Brief Title: Transcutaneous Spinal Cord Stimulation in Healthy Subjects to Activate Central Pattern Generator
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Castilla-La Mancha (Other)
Collaborators: Hospital Nacional de Parapléjicos de Toledo (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: aamg295
Record Dates: First submitted 2020-01-22; First posted 2020-01-27 (Actual); Last update posted 2020-05-01 (Actual); Status verified 2020-04

CONDITIONS: Motor Activity
Keywords: transcutaneous spinal cor stimulation; neuromodulation; motor activity
MeSH Terms: conditions — Motor Activity

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- transcutaneous spinal cord stimulation (Experimental): Transcutaneous application of electrical (biphasic current, 1ms, 30Hz) stimulation over the back for a 10 minutes session.The intensity of the current will increase until motor reflex threshold. If it will not possible, intensity will be increase until participants report a "strong but comfortable" sensation.
  Transcutaneous electrical stimulation over back through the electrotherapy device Myomed 932. (Enraf-Nonius, Delft, Netherlands).
  Interventions: Device: Transcutaneous spinal cord stimulation
- sham stimulation (Experimental): Electrodes are placed over the back for a 10 minutes in the same manner as experimental groups, but will be applied a sham electrical stimulation increasing current intensity during 30 second and decrease intensity subsequently.
  Sham transcutaneous electrical stimulation over back through the electrotherapy device Myomed 932. (Enraf-Nonius, Delft, Netherlands).
  Interventions: Device: Transcutaneous spinal cord stimulation

INTERVENTIONS:
Device: Transcutaneous spinal cord stimulation — Electrodes are placed over the back for a 10 minutes in the same manner as experimental groups, but will be applied a sham electrical stimulation increasing current intensity during 30 second and decrease intensity subsequentl
  Other Names: tSCS

SUMMARY:
The purpose of this study is to determinate whether the application of transcutaneous spinal cord stimulation produce changes in the excitability of alpha moto neurone in healthy volunteers. Moreover evidence whether the effect of the electric currents can increase muscle strength.

DETAILED DESCRIPTION:
In the last years several experimental studies have evidenced that the transcutaneous spinal cord stimulation (tSCS) can evoque spinal reflex activity. The activation of propioceptive afferent would then activated motoneurons innervated at the same metameric and adjacent levels. The possibility of activating neural networks with non-invasive stimulation method opens a therapeutic window for the treatment of different neurological disorders. So the purpose of this study is quantify the modulation of the excitability of alpha motor neurone when the application of the current is in the central nervous system compared with a sham group.

ELIGIBILITY:
Inclusion Criteria:

* Participants will be volunteer healthy students of Physiotherapy, University of Castilla - La Mancha, older than 18 years.

Exclusion Criteria:

* Neuromuscular disease.
* Epilepsy.
* Trauma, surgery or pain affecting the upper limb, shoulder girdle or lumbar área.
* Osteosynthesis material in the upper limb.
* Diabetes.
* Cancer.
* Cardiovascular disease.
* Pacemaker or other implanted electrical device.
* Take any drug (NSAIDs, corticosteroids, antidepressants, analgesics, antiepileptics, ...) during the study and in the previous 7 days.
* Presence of tattoos or other external agent introduced into the treatment or assessment area.
* Pregnancy.
* Sensitivity disturbance in lower limb.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2019-01-30 (Actual); Primary Completion 2020-02-03 (Actual); Study Completion 2020-03-31 (Actual)

PRIMARY OUTCOMES:
Baseline Motor evoked potential (MEP) | baseline at 0 min.
  The action potential elicited by transcranial magnetic stimulation of the motor cortex through the scalp. EMG response will be recorded by surface electrodes (Signa lConditioning Electrodes v2.3, Delsys Inc., USA) fixed in quadriceps and tibialis anterior muscles. by the SENIAM protocol (www.seniam.org).
During treatment Motor evoked potential (MEP) | During treatment at 5 min.
  The action potential elicited by transcranial magnetic stimulation of the motor cortex through the scalp. EMG response will be recorded by surface electrodes (Signa lConditioning Electrodes v2.3, Delsys Inc., USA) fixed in quadriceps and tibialis anterior muscles. by the SENIAM protocol (www.seniam.org).
Post-treatment 1 Motor evoked potential (MEP) | At 2 min after treatment.
  The action potential elicited by transcranial magnetic stimulation of the motor cortex through the scalp. EMG response will be recorded by surface electrodes (Signa lConditioning Electrodes v2.3, Delsys Inc., USA) fixed in quadriceps and tibialis anterior muscles. by the SENIAM protocol (www.seniam.org).
Post-treatment 2 Motor evoked potential (MEP) | At 4 min after treatment.
  The action potential elicited by transcranial magnetic stimulation of the motor cortex through the scalp. EMG response will be recorded by surface electrodes (Signa lConditioning Electrodes v2.3, Delsys Inc., USA) fixed in quadriceps and tibialis anterior muscles. by the SENIAM protocol (www.seniam.org).

SECONDARY OUTCOMES:
Baseline Strength | Baseline at 0 min.
  Hand dynamometer will be used to measure muscle strength. 3 trial of 3 second of isometric muscle contraction of quadriceps and tibialis anterior will be carried.
Post-treatment Strength | At 8 min after treatment.
  Hand dynamometer will be used to measure muscle strength. 3 trial of 3 second of isometric muscle contraction of quadriceps and tibialis anterior will be carried.

CONTACTS AND LOCATIONS:
Overall Officials: Julio Gómez-Soriano, PhD, Principal Investigator — Castilla-La Mancha University
Locations (3):
- Spain (3):
  - Julio, Toledo
  - Álvaro, Toledo
  - Diego Serrano-Muñoz, Toledo

IPD SHARING:
Plan to Share IPD: No